CLINICAL TRIAL: NCT02669602
Title: Dynamic Mediterranean Prospective Cohort: the SUN Project
Status: Enrolling by invitation | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: SUN
Record Dates: First submitted 2016-01-11; First posted 2016-02-01 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Lifestyle; Chronic Disease; Dietary Habits
Keywords: Nutritional epidemiology; Prospective
MeSH Terms: conditions — Chronic Disease; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No intervention: No Intervention

SUMMARY:
Dynamic prospective cohort of Spanish university graduates. The main objective is to evaluate the associations between nutrition and lifestyle and chronic diseases.

DETAILED DESCRIPTION:
The SUN Project (University of Navarra Follow-Up Study) began in 1999, and currently more than 20,500 people participate. The Project is permanently open to new volunteers, and around 2,000 new participants are invited each year.

A new questionnaire is sent to participants every two years. The questionnaires are named with the letter "Q," followed by the number of years that have passed since the participant first volunteered. The first questionnaire is titled "Q0" and is followed by "Q2","Q4", etc.

The cohort is "dynamic" thanks to the fact that it is permanently open to new volunteers. Although the Project was created by the Department of Preventive Medicine and Public Health of the University of Navarra, it now counts on the invaluable collaboration of other Spanish university centers.

Thanks to the invaluable collaboration of our participants, the investigators are able to research cardiovascular diseases, depression, fertility, arterial hypertension, and car accident injuries, among other areas.

ELIGIBILITY:
Inclusion Criteria:

* Spanish university graduates

Exclusion Criteria:

* not Spanish university graduates

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Spanish university graduates
Sampling Method: Non-Probability Sample
Enrollment: 22500 (Estimated)
Dates: Start 1999-12 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2075-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 50 years

SECONDARY OUTCOMES:
Cardiovascular disease | 50 years
  cardiovascular death, acute coronary syndromes (myocardial infarction with or without ST elevation), revascularization procedures or fatal or non-fatal stroke.
Obesity | 50 years
  BMI>30 kg/m2
Depression | 50 years
  Diagnosed depression through the Structured Clinical Interview (SCID-I) for the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
Cognitive function | 50 years
  Telephone Interview of Cognitive Status-modified (TICS-m)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Martinez-Gonzalez, PhD, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Carlos S, De La Fuente-Arrillaga C, Bes-Rastrollo M, Razquin C, Rico-Campa A, Martinez-Gonzalez MA, Ruiz-Canela M. Mediterranean Diet and Health Outcomes in the SUN Cohort. Nutrients. 2018 Mar 31;10(4):439. doi: 10.3390/nu10040439. PMID 29614726
- [Result] Segui-Gomez M, de la Fuente C, Vazquez Z, de Irala J, Martinez-Gonzalez MA. Cohort profile: the 'Seguimiento Universidad de Navarra' (SUN) study. Int J Epidemiol. 2006 Dec;35(6):1417-22. doi: 10.1093/ije/dyl223. Epub 2006 Oct 22. No abstract available. PMID 17060332
- [Derived] de la O V, Goni L, Zazpe I, Martinez-Gonzalez MA, Santiago S, Bes-Rastrollo M, Ruiz-Canela M. Long-term risk of overweight/obesity according to the protein quality index in a prospective middle-aged cohort. Clin Nutr. 2025 Sep;52:284-298. doi: 10.1016/j.clnu.2025.07.024. Epub 2025 Jul 30. PMID 40816209
- [Derived] Gribble AK, Hershey MS, Lopez-Gil JF, Lan FY, Kales SN, Martinez-Gonzalez MA, Bes-Rastrollo M, Fernandez-Montero A. Role of the Intensity of Habitual Physical Activity in the Maintenance of Normal Blood Pressure: Findings From the SUN Longitudinal Cohort Study. J Am Heart Assoc. 2025 Jun 17;14(12):e038664. doi: 10.1161/JAHA.124.038664. Epub 2025 Jun 5. PMID 40470663
- [Derived] Martinez-Gonzalez MA. Should we remove wine from the Mediterranean diet?: a narrative review. Am J Clin Nutr. 2024 Feb;119(2):262-270. doi: 10.1016/j.ajcnut.2023.12.020. Epub 2023 Dec 28. PMID 38157987
- [Derived] Talavera-Rodriguez I, Fernandez-Lazaro CI, Hernandez-Ruiz A, Hershey MS, Galarregui C, Sotos-Prieto M, de la Fuente-Arrillaga C, Martinez-Gonzalez MA, Ruiz-Canela M. Association between an oxidative balance score and mortality: a prospective analysis in the SUN cohort. Eur J Nutr. 2023 Jun;62(4):1667-1680. doi: 10.1007/s00394-023-03099-8. Epub 2023 Feb 12. PMID 36781422
- [Derived] Bazal P, Gea A, Navarro AM, Salas-Salvado J, Corella D, Alonso-Gomez A, Fito M, Munoz-Bravo C, Estruch R, Fiol M, Lapetra J, Serra-Majem L, Ros E, Rekondo J, Munoz MA, Basora J, Sorli JV, Toledo E, Martinez-Gonzalez MA, Ruiz-Canela M. Caffeinated coffee consumption and risk of atrial fibrillation in two Spanish cohorts. Eur J Prev Cardiol. 2021 May 22;28(6):648-657. doi: 10.1177/2047487320909065. PMID 34021573
- [Derived] Alonso-Pedrero L, Ojeda-Rodriguez A, Zalba G, Razquin C, Martinez-Gonzalez MA, Bes-Rastrollo M, Marti A. Association between ideal cardiovascular health and telomere length in participants older than 55 years old from the SUN cohort. Rev Esp Cardiol (Engl Ed). 2022 Apr;75(4):308-315. doi: 10.1016/j.rec.2021.04.002. Epub 2021 May 14. English, Spanish. PMID 33994338
- [Derived] Martin-Calvo N, Santiago Neri S, Segura G, Fernandez-Lazaro CI, Barberia-Latasa M, Martinez-Gonzalez MA. Pregestational BMI and higher offspring's risk of overweight/obesity in smoker and non-smoker mothers. Public Health Nutr. 2021 Sep;24(13):4204-4211. doi: 10.1017/S1368980020005194. Epub 2020 Dec 18. PMID 33336642
- [Derived] Hershey MS, Fernandez-Montero A, Sotos-Prieto M, Kales S, Gea A, Ruiz-Estigarribia L, Sanchez-Villegas A, Diaz-Gutierrez J, Martinez-Gonzalez MA, Ruiz-Canela M. The Association Between the Mediterranean Lifestyle Index and All-Cause Mortality in the Seguimiento Universidad de Navarra Cohort. Am J Prev Med. 2020 Dec;59(6):e239-e248. doi: 10.1016/j.amepre.2020.06.014. Epub 2020 Nov 18. PMID 33220762
- [Derived] Alonso-Pedrero L, Ojeda-Rodriguez A, Martinez-Gonzalez MA, Zalba G, Bes-Rastrollo M, Marti A. Ultra-processed food consumption and the risk of short telomeres in an elderly population of the Seguimiento Universidad de Navarra (SUN) Project. Am J Clin Nutr. 2020 Jun 1;111(6):1259-1266. doi: 10.1093/ajcn/nqaa075. PMID 32330232
- [Derived] Gardeazabal I, Romanos-Nanclares A, Martinez-Gonzalez MA, Castello A, Sanchez-Bayona R, Perez-Gomez B, Razquin C, Aramendia-Beitia JM, Pollan M, Toledo E. Mediterranean dietary pattern is associated with lower incidence of premenopausal breast cancer in the Seguimiento Universidad de Navarra (SUN) Project. Public Health Nutr. 2020 Dec;23(17):3148-3159. doi: 10.1017/S1368980019003835. Epub 2020 Feb 24. PMID 32090723
- [Derived] Rico-Campa A, Martinez-Gonzalez MA, Alvarez-Alvarez I, Mendonca RD, de la Fuente-Arrillaga C, Gomez-Donoso C, Bes-Rastrollo M. Association between consumption of ultra-processed foods and all cause mortality: SUN prospective cohort study. BMJ. 2019 May 29;365:l1949. doi: 10.1136/bmj.l1949. PMID 31142450
- [Derived] Fresan U, Martinez-Gonzalez MA, Sabate J, Bes-Rastrollo M. Global sustainability (health, environment and monetary costs) of three dietary patterns: results from a Spanish cohort (the SUN project). BMJ Open. 2019 Feb 21;9(2):e021541. doi: 10.1136/bmjopen-2018-021541. PMID 30796113
- [Derived] Garcia-Arellano A, Martinez-Gonzalez MA, Ramallal R, Salas-Salvado J, Hebert JR, Corella D, Shivappa N, Forga L, Schroder H, Munoz-Bravo C, Estruch R, Fiol M, Lapetra J, Serra-Majem L, Ros E, Rekondo J, Toledo E, Razquin C, Ruiz-Canela M; SUN and PREDIMED Study Investigators. Dietary inflammatory index and all-cause mortality in large cohorts: The SUN and PREDIMED studies. Clin Nutr. 2019 Jun;38(3):1221-1231. doi: 10.1016/j.clnu.2018.05.003. Epub 2018 May 24. PMID 30651193
- [Derived] Mendonca RD, Carvalho NC, Martin-Moreno JM, Pimenta AM, Lopes ACS, Gea A, Martinez-Gonzalez MA, Bes-Rastrollo M. Total polyphenol intake, polyphenol subtypes and incidence of cardiovascular disease: The SUN cohort study. Nutr Metab Cardiovasc Dis. 2019 Jan;29(1):69-78. doi: 10.1016/j.numecd.2018.09.012. Epub 2018 Oct 4. PMID 30459074
- [Derived] Mendonca RD, Pimenta AM, Gea A, de la Fuente-Arrillaga C, Martinez-Gonzalez MA, Lopes AC, Bes-Rastrollo M. Ultraprocessed food consumption and risk of overweight and obesity: the University of Navarra Follow-Up (SUN) cohort study. Am J Clin Nutr. 2016 Nov;104(5):1433-1440. doi: 10.3945/ajcn.116.135004. Epub 2016 Oct 12. PMID 27733404
- See also: Web page of the SUN cohort — https://www.unav.edu/web/departamento-de-medicina-preventiva-y-salud-publica/proyecto-sun